CLINICAL TRIAL: NCT02347449
Title: The Impact of the Oncotype DX® Breast Cancer Assay on Treatment Decisions in a Canadian Population of Patients With Estrogen Receptor- Positive Early Breast Cancer With 1-3 Positive Lymph Nodes
Brief Title: The Impact of the Oncotype DX® Breast Cancer Assay on Treatment Decisions in a Canadian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 231-2014
Record Dates: First submitted 2014-11-17; First posted 2015-01-27 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast
Keywords: Early-stage Breast cancer, node positive; Prognosis; Oncotype Dx
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early stage breast cancer (Experimental): Women with node positive (1-3 nodes), ER positive breast cancer who are receiving (or will receive) endocrine therapy, and who are candidates for chemotherapy.
  Study subjects will have ONCOTYPE Dx assay performed on their breast tumors, and will complete study questionnaires.
  Interventions: Other: Questionnaires, Oncotype Dx Assay

INTERVENTIONS:
Other: Questionnaires, Oncotype Dx Assay — 1. Physician pre-assay questionnaire
  2. Patient pre-assay questionnaire
  3. Oncotype DX® Assay
  4. Physician post- assay questionnaire
  5. Patient post-assay questionnaire
  Other Names: Oncotype Dx Assay, Questionnaires

SUMMARY:
The main goal of this study is to characterize whether the results of the Oncotype DX® assay affect the physician's treatment recommendations for the adjuvant treatment of women with ER-positive (ER+), early breast cancer (EBC) with 1-3 positive lymph nodes who are potential candidates for chemotherapy, but for whom the benefits of chemotherapy may be uncertain.

DETAILED DESCRIPTION:
The Oncotype DX assay has been commercially available in the U.S. since 2004 as a tool to aid a physician's treatment recommendation for a breast cancer patient. While the Oncotype DX assay is currently reimbursed by the Ontario Health Ministry for node-negative EBC, it is not reimbursed for node-positive (N+) patients although the assay has been shown to be both prognostic and predictive of chemotherapy benefit for patients with N+ disease.

The goal of this study is to characterize how the results of the Oncotype DX® assay impact the decision making processes of physicians and patients in a large academic medical center in Ontario by evaluating recommendations for adjuvant therapy within a population of ER+, N+ EBC patients with 1 to 3 positive lymph nodes for whom the benefit of adjuvant chemotherapy is not certain.

Upon consent, the patient will be assigned an ID number. The physician will discuss the patient's treatment alternatives prior to ordering the Oncotype DX assay. After discussion with the patient, the physician will complete a baseline questionnaire indicating the therapeutic strategy he/she would recommend to the patient based upon the available clinical and pathologic data. In addition, the patient will also complete a baseline questionnaire indicating her treatment preference, based on the previous discussion with the physician.

The Oncotype DX assay will be ordered after receipt of the Registration and Confirmation of Eligibility Form and assignment of patient study number. Once the results of the Oncotype DX assay are available, the physician will discuss the results with the patient. Both the physician and the patient will complete separate follow-up post-assay questionnaires after the results of the Oncotype DX assay are known and shared with the patient.

One last form completed by a study manager or coordinator after a treatment plan has been initiated will register the actual treatment administered to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have undergone surgical treatment for breast cancer with adequate evaluation of lymph node status with a sentinel lymph node procedure or full axillary dissection, with positive involvement of 1-3 axillary lymph nodes as confirmed by histologic examination.
* ECOG performance status 0 or 1
* Patient must be a candidate for treatment of their cancer with systemic chemotherapy in addition to hormonal therapy
* Eligible Staging Criteria: T1-3 N1 M0
* Breast tumor must undergo central pathology review at GHI and must be found adequate for the Oncotype DX assay.
* Breast tumor must be estrogen-receptor positive and HER2 positive (IHC/FISH) as per institutional guidelines

Exclusion Criteria:

* Patient has a prior history of breast cancer in the same breast
* Patient as been newly diagnosed with more than one operable primary breast tumor
* Patient has multi-centric tumors (note: patients with multi-focal tumors may be included)
* Patient has known metastatic breast cancer
* Patient has <2mm invasive tumor as assessed by local pathologist
* Patient has received any kind of neoadjuvant treatment
* Presence of clinical factors rendering the patient a non-viable candidate for adjuvant chemotherapy
* Presence of a current medical condition that would interfere with patient's ability to consent and participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Change in physicians' treatment recommendations | 2-4 weeks

SECONDARY OUTCOMES:
Change in patient's treatment preference and level of confidence in treatment plan | 2-4 weeks
Change in physicians' level of confidence in the treatment recommendation | 2-4 weeks
Specific chemotherapy and/or hormone therapy regimen received by patient | 4-8 weeks
  Assessment of actual adjuvant treatment given to patient after Oncotype DX results available

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Eisen, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada